CLINICAL TRIAL: NCT05674162
Title: Observer Reactivity During Gait Measurements in a Clinical Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sint Maartenskliniek (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1042_TZO_Observer Reactivity
Record Dates: First submitted 2022-12-21; First posted 2023-01-06 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2022-12

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — No-Observed-Adverse-Effect Level

STUDY DESIGN:
Intervention Model Description: Single group, repeated measures model.
Masking Description: The participants are masked to existence of different conditions, not to the measurement of their data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gait measurement (Experimental): Use of four accellerometers/sensors (1 on each foot, one on the lumbar area and one on the sternum) that measure gait parameters during walking.
  Interventions: Behavioral: Unobserved; Behavioral: Observed; Radiation: Unobserved & Measured

INTERVENTIONS:
Behavioral: Unobserved — Participants walk a distance of 40 meters wearing the sensors, unobserved by the researcher.
Behavioral: Observed — Participants walk a distance of 40 meters wearing the sensors, observed by the researcher.
Radiation: Unobserved & Measured — Participants walk a distance of 40 meters wearing the sensors, unobserved by the researcher and aware of the gait measurement by the sensors.

SUMMARY:
Observer reactivity, also known as the 'Hawthorne effect', can roughly be described as the alteration of behaviour as a consequence of observation or awareness of measurement. Although researchers are aware of a potential observation effect during measurements, observer reactivity may also influence assessments that are performed as part of clinical care. Previous research on observer reactivity during gait measurements has resulted in contradicting outcomes and most studies examined the effects of participation in research rather than the clinical measurement of gait in a gait lab setting or the observation by professionals. Therefore, the aim of this study is to examine the differences in gait pattern between unobserved walking, observed walking, and observed walking combined with awareness of measurement, in a within-subjects repeated measures design.

DETAILED DESCRIPTION:
Observer reactivity, also known as the 'Hawthorne effect', can roughly be described as the alteration in behaviour as a consequence of observation or awareness of measurement. It is believed that this could influence research outcomes in prospective experimental and observational studies. However, as described in a recent systematic review, the extend of the effect on research outcomes is still debated. The available studies on observer reactivity with various populations and tasks generate contradicting findings and conclusions. Especially within the health sciences, more research is necessary as observer reactivity may confound study results in the direction of better health outcomes.

Previous research on observer reactivity during gait measurements has resulted in contradicting outcomes. For example, some studies showed a higher walking velocity and better gait symmetry under observation, while others showed an opposite effect. This may be caused by the variation in diagnosis group between the studies or small sample sizes. Because of these mixed results and the low number of studies available on this topic, there is yet no consensus on a generalizable effect of observation during gait measurements. Furthermore, most studies examine the effects of participation in research rather than the clinical measurement of gait in a gait lab setting or the observation by professionals.

For clinical decision making, it is essential to investigate whether gait measurements are representative for the actual gait pattern of the patient. Therefore, the aim of this study is to examine the differences in gait pattern between unobserved walking, observed walking by a researcher, and observed walking combined with awareness of measurement by sensors.

ELIGIBILITY:
Inclusion Criteria:

* Subacute or chronic stroke (>3 months ago)

Exclusion Criteria:

* Not able to walk 50 meters without resting.
* Not able to understand instructions given by the researcher.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Gait velocity | 5 minutes
  Mean walking speed (meters/second)

SECONDARY OUTCOMES:
Stride length | 5 minutes
  Mean stride length (meters)
Cadance | 5 minutes
  Cadance (steps/minute)
Stance time symmetry | 5 minutes
  Symmetry in stance time between paretic and non-paretic leg
Swing time symmetry | 5 minutes
  Symmetry in swing time between paretic and non-paretic leg
percent single leg stance | 5 minutes
  percent single leg stance of the total gait cycle of the paretic leg
percent single leg stance symmetry | 5 minutes
  Symmetry in percent single leg stance between paretic and non-paretic leg
Stride length variability | 5 minutes
  Variability in stride length
Swing time variability | 5 minutes
  Variability in swing time of the paretic leg

OTHER OUTCOMES:
Fugl Meyer Assessment of Lower Extremities | 2 minutes
  Stages 3 and 4, both ranging from minimum 0 to maximum 4 points, with a higher score meaning a better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Noël LW Keijsers, PhD, Principal Investigator — Sint Maartenskliniek
Locations (1):
- Sint Maartenskliniek, Ubbergen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No